CLINICAL TRIAL: NCT06249750
Title: Clinical Application of Near-infrared Whole Body Heat Shock Multimodal Technique in Treatment of Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pengyuan Liu (Other)
Responsible Party: Sponsor-Investigator, Pengyuan Liu, Research Secretary, Zhejiang Hospital
Organization: Zhejiang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEAIS007
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (CRPC)
Keywords: hyperthermia, immune checkpoint inhibitor, RTK inhibitor, CRPC
MeSH Terms: conditions — Hyperthermia | interventions — Immunotherapy; Immune Checkpoint Inhibitors; tislelizumab; anlotinib; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immuno-targeted therapy group (Experimental): ICI regimen: Tislelizumab, 200mg, ivgtt., d1, q21d; RTK inhibitor regimen: Anlotinib, 12mg (at an initial dose of 12mg, later adjusted according to the instructions), po., d1~14, q21d.
  Interventions: Drug: Immunotherapy; Drug: Targeted therapy
- Hyperthermia-immuno-targeted therapy group (Experimental): ET-SPACE near-infrared irradiation whole-body hyperthermia: d1, d8, q21d, rectal temperature reaches 38.5~39 ℃ and then maintain 1h. ICI regimen: Tislelizumab, 200mg, ivgtt., d2, q21d; RTK inhibitor regimen: Anlotinib, 12mg (at an initial dose of 12mg, later adjusted according to the instructions), po., d2~15, q21d.
  Interventions: Drug: Immunotherapy; Drug: Targeted therapy; Device: Hyperthermia

INTERVENTIONS:
Drug: Immunotherapy — Immunotherapy is currently a hot spot in the field of tumor research. Immune Checkpoint Inhibitor (ICI) is a monoclonal antibody designed to target the negative immunoregulatory pathway overexpressed in tumor cells, which can release the anti-tumor immunosuppressive signals and restore the killing of tumors by the immune cells, and thus exert anti-tumor effects. ICI regimen: Tislelizumab, 200mg, ivgtt., d1, q21d.
  Other Names: Immune checkpoint inhibitor; ICI; Tislelizumab (BeiGene, China)
Drug: Targeted therapy — Recent studies have found that the combination of RTK inhibitors and ICIs can exert synergistic effects on different mechanisms, which can compensate for the deficiencies of single-agent RTK inhibitors and single-agent ICIs in the treatment of CRPC and become a potential novel therapeutic strategy for solid malignant tumors. RTK inhibitor regimen: Anlotinib, 12mg, po., d2~15, q21d.
  Other Names: RTK inhibitor; Anlotinib (CHIATAI TIANQING PHARMACEUTICAL GROUP, China)
Device: Hyperthermia — Thermal stimulation is a rapidly developing physiotherapeutic tool, which is playing an increasingly important role in the field of comprehensive tumor therapy due to its unique low adverse effects and high compatibility. A large number of clinical studies have shown that the addition of heat stress to multimodal tumor therapy does not significantly increase toxicity and side effects, and the combination of heat stress with other therapies can have the effect of "1+1>2". ET-SPACE near-infrared irradiation whole-body hyperthermia: d1, d8, q21d, rectal temperature reaches 38.5~39 ℃ and then maintain 1h.
  Other Names: ET-SPACE whole body hyperthermia; near infrared irradiation; ET-SPACE™ (Shenzhen ET medical, China); heat stress
  Arms: Hyperthermia-immuno-targeted therapy group

SUMMARY:
In this study, we propose to use the combination of ET-SPACE NIR irradiation whole-body thermal stimulation, ICI (Tislelizumab), and RTK inhibitor (Anlotinib) in the multimodal treatment of CRPC.

DETAILED DESCRIPTION:
The initial efficacy and safety of the multimodal therapy will be evaluated at the animal level to fully validate the potential feasibility of the therapy. Subsequently, the efficacy of the multimodal therapy will be verified at the organoid level, and based on which a translational randomized controlled clinical trial will be conducted to evaluate the efficacy and safety of the multimodal therapy at the human level, and the patients will be followed up for a long period of time, so as to collect detailed data on improvement of the quality of life. Finally, the synergistic effect of the multimodal therapy will be analyzed at the molecular and cellular levels.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of PC and clinically confirmed diagnosis of CRPC;
* Complete and reliable medical history and medical records;
* No other primary tumors except CRPC;
* Blood tests, liver function, renal function and electrocardiogram are basically normal;
* Patients with ECOG score 0~3, aged ≥18 years and <90 years old;
* Patients with good compliance, able to accept regular follow-up.

Exclusion Criteria:

* History of malignant tumor other than PC within the past 5 years;
* Severe abnormalities in the patient's laboratory indices may jeopardize patient safety or compromise this study;
* Accompanied by severe underlying diseases that cannot tolerate this therapy;
* With acute diseases, such as acute infection, active bleeding;
* Those who have recently participated in other clinical trials and have not passed the washout period;
* Those who cannot tolerate systemic heat stress, such as claustrophobic patients;
* Those who have a history of allergy to the drugs used in the trial;
* Patients with other reasons for not being able to be enrolled in the study, according to the study doctor.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical objective response rate (BORR) | 3 weeks
  Detect blood PSA levels before and during treatment, compare baseline and post treatment PSA difference levels, and evaluate efficacy.
  Bio Complete Response (BCR): PSA remains normal or decreases to normal (4ng/mL) for at least 3 weeks.
  Partial Biochemical Response (BPR): PSA decreased by ≥ 50% from baseline and maintained for at least 3 weeks.
  BPRR=BCR+BPR/All patients × 100%.

SECONDARY OUTCOMES:
Bio-Disease Control Rate （BDCR） | 3 weeks
  Bio Complete Response (BCR): PSA remains normal or decreases to normal (4ng/mL) for at least 3 weeks.
  Partial Biochemical Response (BPR): PSA decreased by ≥ 50% from baseline and maintained for at least 3 weeks.
  Bio Progression Disease (BPD): PSA increased by ≥ 25% from baseline. BDCR=BCR+BPR+BPD/All patients × 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No